CLINICAL TRIAL: NCT06909864
Title: Competitive Swimming and Shoulder Adaptations: The Role of Stroke Specialty in Adolescent Swimmers
Acronym: Shoulder
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERCAN YILLI, Clinical Physical Therapist, Hacettepe University
Other Study IDs: GO 19/823
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Swimming; Shoulder; Adolescent
Keywords: Swimming; Shoulder; Adolescent; Musculoskeletal screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Swimming Group (SWG): The asymptomatic swimmers with no history of major upper limb injury or surgery and no injury history of upper limb in last 6 months, having experience in at least 5 years competitive swimming, actively participating in competitive swimming at least 1 year, competing at least in national level and having swimming stroke specialization in competitive swimming were included
- Control Group (CG): The non-athlete peers with no competed in overhead sports like swimming, basketball, volleyball, tennis, baseball as professional or recreational, no history of major upper limb injury or surgery and no injury history in last 6 months participated in this study.

SUMMARY:
Objectives: To examine the sport-specific adaptations and investigate the effect of swimming stroke specialization in shoulder complex among adolescent competitive swimmers.

Design: Observational study.

Setting: Athletic facilities.

Participants: A total of 76 adolescents participated including n = 28 non-swimmers as Control Group (CG) and n = 48 competitive swimmers as Swimmers Group (SWG).

Main Outcome Measures: Strength of glenohumeral (GH) and scapular muscles (SM), mobility of GH (GH ROMs) joint, proprioception, pectoralis minor length (PML), posterior shoulder tightness (PST) were evaluated for all participants. Kerlan Jobe Orthopaedic Score (KJOC) was sed to evaluate for SWG. The tested shoulder physical performance parameters were compared between the groups.

ELIGIBILITY:
Inclusion Criteria for Swimmer Group:

* aged between 13 to 18 years
* the asymptomatic swimmers with no history of major upper limb injury or surgery and no injury history of upper limb in last 6 months
* having experience in at least 5 years competitive swimming,
* actively participating in competitive swimming at least 1 year,
* competing at least in national level and having swimming stroke specialization in competitive swimming

Inclusion Criteria for Control Group:

* aged between 13 to 18 years,
* no competed in overhead sports like swimming, basketball, volleyball, tennis, baseball as professional or recreational,
* no history of major upper limb injury or surgery in last 6 months.

Exclusion Criteria for all participants:

* if they had at least two positive signs by shoulder screening tests (Hawkin's/Kennedy Subacromial Impingement Test, Jobe/Empty Can Test, External Rotation Resistance Test, Apprehension Instability Test, Speed Test and Gerber Lift-Off Test),
* a BMI of 30 kg/m² or greater than 30 kg/m²,
* competing in paralympic sports,
* if they had any major upper limb injuries or surgeries,
* if they had any systemic, neurological or rheumatological diseases,
* being pre-pubertal stage (Tanner I) according to Tanner Scale,
* indicated their unwillingness to participate to this study.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 55 adolescent competitive swimmers and 40 non-athlete peers were screened. 48 swimmers and 28 non-athlete peers aged between 13 to 18 years met the inclusion criteria and participated in this study
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | From October 2019 to September 2021
  Muscle strength was assessed with break test by using hand-hold dynamometer (Jamaar Hand Dynamometer, USA). Assessments were applied for both shoulders and 3 times for each position. Shoulder flexion, extension, abduction, full-can, glenohumeral IR and ER, upper, middle and lower trapezius, serratus anterior muscle tests were applied. GH ER/IR ratio was calculated as well (21-26). Measurements were recorded in Newton (N).
Range of Motion | From October 2019 to September 2021
  Passive Range of Motion (PROM) of both shoulders was assessed using a digital inclinometer (Get My ROM, version 1.0.3 for iOS; Interactive Medical Productions, Hampton, NH, USA). Shoulder internal rotation (IR), external rotation (ER), and total-rotational ROM were assessed (ICC = 0.92-94). Shoulder IR and ER PROM were obtained with the participant lying supine on a standard examination table, with the shoulder initially abducted to 90° with 0° rotation and the elbow flexed to 90° with neutral pronation/supination. In addition, Total-rotational ROM was calculated by summing the IR and ER ROMs average degrees of each shoulder.
Pectoralis Minor Length | From October 2019 to September 2021
  Digitized 2 anatomical landmarks representing the length of the pectoralis minor. These 2 points were the medial-inferior angle of the coracoid process and just lateral to the sternocostal junction of the inferior aspect of the fourth rib. Measurements of pectoralis minor muscle length was taken with tape measure (ICC = 0.96). Because of height and muscle length variability among subjects, a normalization index was developed. The pectoralis minor index (PMI) was calculated by dividing the resting muscle length measurement by the subject height and multiplying by 100.
Proprioception | From October 2019 to September 2021
  For proprioception testing, participants attempted to reproduce 45° ER angle. Participants were positioned as lying supine with arm abducted to 90°, elbow flexed at 90°. The ''Get My ROM'' digital inclinometer was used to measure the angles; the iPhone was securely attached to participants forearm using a strap with the screen facing the tester (ICC = 0.87-89). The participant was instructed to close their eyes by using an eye patch throughout testing. The arm was passively rotated to 45° ER and held in this position for 3 seconds. The participant was asked to remember this position. Following the return to neutral the participant was asked to actively return the arm back to the angle shown. The amount of degrees away from 45° was recorded.
Posterior Shoulder Tightness | From October 2019 to September 2021
  Participants were positioned supine with both shoulders flush against a standard examination table. The tester stood at the head of the examination table toward the head of the subject and positioned the test shoulder and elbow in 90 of both abduction and flexion. To measure GH horizontal adduction, The ''Get My ROM'' digital inclinometer was aligned with the ventral midline of the humerus. The angle created by the end position of the humerus with respect to 0 of horizontal adduction was then recorded as the total amount of GH horizontal adduction motion (ICC = 0.79).

SECONDARY OUTCOMES:
Scapular Dyskinesis | From October 2019 to September 2021
  Each participant performed 5 repetitions of bilateral, active, weighted shoulder flexion and bilateral, active, weighted shoulder abduction (frontal plane) while they were observed from the posterior views. First of all, the scapula was observed while participants in rest and then weighted shoulder flexion and abduction movements from the posterior views. Kibler et al. reported the reliability of a visually based classification system for scapular dysfunction that defined 3 different types of motion abnormalities: Type 1 = inferior angle prominence, Type II = medial border prominence and Type III = excessive superior border elevation. Normal, symmetric scapular motion was considered Type IV (ICC = 0.32-42).
Kerlan-Jobe Orthopaedic Clinic Shoulder and Elbow Score (KJOC) | From October 2019 to September 2021
  KJOC has been designed specifically as a subjective assessment tool to measure functional status of the upper extremities in overhead athletes. The KJOC was translated from English to Turkish to enable use of questionnaires in Turkish overhead athletes by Turgut et al. KJOC was used to measure functional status of the upper extremities in competitive adolescent swimmers and the scores compared in different stroke specialty among the swimmers in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Cebeci Sports Complex, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laudner KG, Stanek JM, Meister K. Assessing posterior shoulder contracture: the reliability and validity of measuring glenohumeral joint horizontal adduction. J Athl Train. 2006 Oct-Dec;41(4):375-80. PMID 17273461
- [Background] Kibler WB, McMullen J. Scapular dyskinesis and its relation to shoulder pain. J Am Acad Orthop Surg. 2003 Mar-Apr;11(2):142-51. doi: 10.5435/00124635-200303000-00008. PMID 12670140
- [Background] McClure P, Tate AR, Kareha S, Irwin D, Zlupko E. A clinical method for identifying scapular dyskinesis, part 1: reliability. J Athl Train. 2009 Mar-Apr;44(2):160-4. doi: 10.4085/1062-6050-44.2.160. PMID 19295960
- [Background] Higson E, Herrington L, Butler C, Horsley I. The short-term effect of swimming training load on shoulder rotational range of motion, shoulder joint position sense and pectoralis minor length. Shoulder Elbow. 2018 Oct;10(4):285-291. doi: 10.1177/1758573218773539. Epub 2018 May 12. PMID 30214495
- [Background] Ager AL, Roy JS, Roos M, Belley AF, Cools A, Hebert LJ. Shoulder proprioception: How is it measured and is it reliable? A systematic review. J Hand Ther. 2017 Apr-Jun;30(2):221-231. doi: 10.1016/j.jht.2017.05.003. PMID 28641738
- [Background] Robertson JA. F. P. Kendall and E. K. McCreary "Muscles, Testing and Function" (Third Edition). Br J Sports Med. 1984;18(1):25-.
- [Background] Michener LA, Boardman ND, Pidcoe PE, Frith AM. Scapular muscle tests in subjects with shoulder pain and functional loss: reliability and construct validity. Phys Ther. 2005 Nov;85(11):1128-38. PMID 16253043
- [Background] Hislop H, Avers D, Brown M. Daniels and Worthingham's muscle Testing-E-Book: Techniques of manual examination and performance testing: Elsevier Health Sciences; 2013.
- [Background] Itoi E, Kido T, Sano A, Urayama M, Sato K. Which is more useful, the "full can test" or the "empty can test," in detecting the torn supraspinatus tendon? Am J Sports Med. 1999 Jan-Feb;27(1):65-8. doi: 10.1177/03635465990270011901. PMID 9934421
- [Background] Hayes K, Walton JR, Szomor ZL, Murrell GA. Reliability of 3 methods for assessing shoulder strength. J Shoulder Elbow Surg. 2002 Jan-Feb;11(1):33-9. doi: 10.1067/mse.2002.119852. PMID 11845146
- [Background] McLaine SJ, Ginn KA, Fell JW, Bird ML. Isometric shoulder strength in young swimmers. J Sci Med Sport. 2018 Jan;21(1):35-39. doi: 10.1016/j.jsams.2017.05.003. Epub 2017 May 25. PMID 28844605
- [Background] Harput G, Guney H, Toprak U, Kaya T, Colakoglu FF, Baltaci G. Shoulder-Rotator Strength, Range of Motion, and Acromiohumeral Distance in Asymptomatic Adolescent Volleyball Attackers. J Athl Train. 2016 Sep;51(9):733-738. doi: 10.4085/1062-6050-51.12.04. Epub 2016 Nov 4. PMID 27813683
- [Background] Rose MB, Noonan T. Glenohumeral internal rotation deficit in throwing athletes: current perspectives. Open Access J Sports Med. 2018 Mar 19;9:69-78. doi: 10.2147/OAJSM.S138975. eCollection 2018. PMID 29593438
- [Background] Wymore L, Reeve RE, Chaput CD. No correlation between stroke specialty and rate of shoulder pain in NCAA men swimmers. Int J Shoulder Surg. 2012 Jul;6(3):71-5. doi: 10.4103/0973-6042.102555. PMID 23204760
- [Background] Park HB, Yokota A, Gill HS, El Rassi G, McFarland EG. Diagnostic accuracy of clinical tests for the different degrees of subacromial impingement syndrome. J Bone Joint Surg Am. 2005 Jul;87(7):1446-55. doi: 10.2106/JBJS.D.02335. PMID 15995110
- [Background] Drigny J, Gauthier A, Reboursiere E, Guermont H, Gremeaux V, Edouard P. Shoulder Muscle Imbalance as a Risk for Shoulder Injury in Elite Adolescent Swimmers: A Prospective Study. J Hum Kinet. 2020 Oct 31;75:103-113. doi: 10.2478/hukin-2020-0041. eCollection 2020 Oct. PMID 33312299
- [Background] Evershed J, Burkett B, Mellifont R. Musculoskeletal screening to detect asymmetry in swimming. Phys Ther Sport. 2014 Feb;15(1):33-8. doi: 10.1016/j.ptsp.2013.02.002. Epub 2013 May 20. PMID 23702323
- [Background] Wanivenhaus F, Fox AJ, Chaudhury S, Rodeo SA. Epidemiology of injuries and prevention strategies in competitive swimmers. Sports Health. 2012 May;4(3):246-51. doi: 10.1177/1941738112442132. PMID 23016094
- [Background] Davis DD, Nickerson M, Varacallo MA. Swimmer's Shoulder. 2023 Nov 22. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470589/ PMID 29262079
- [Background] De Martino I, Rodeo SA. The Swimmer's Shoulder: Multi-directional Instability. Curr Rev Musculoskelet Med. 2018 Jun;11(2):167-171. doi: 10.1007/s12178-018-9485-0. PMID 29679207
- [Background] Aspenes S, Kjendlie PL, Hoff J, Helgerud J. Combined strength and endurance training in competitive swimmers. J Sports Sci Med. 2009 Sep 1;8(3):357-65. eCollection 2009. PMID 24149998
- [Background] Tate A, Turner GN, Knab SE, Jorgensen C, Strittmatter A, Michener LA. Risk factors associated with shoulder pain and disability across the lifespan of competitive swimmers. J Athl Train. 2012 Mar-Apr;47(2):149-58. doi: 10.4085/1062-6050-47.2.149. PMID 22488280
- [Background] Hibberd EE, Myers JB. Practice habits and attitudes and behaviors concerning shoulder pain in high school competitive club swimmers. Clin J Sport Med. 2013 Nov;23(6):450-5. doi: 10.1097/JSM.0b013e31829aa8ff. PMID 24042443
- [Background] Heinlein SA, Cosgarea AJ. Biomechanical Considerations in the Competitive Swimmer's Shoulder. Sports Health. 2010 Nov;2(6):519-25. doi: 10.1177/1941738110377611. PMID 23015983
- [Background] Walker H, Gabbe B, Wajswelner H, Blanch P, Bennell K. Shoulder pain in swimmers: a 12-month prospective cohort study of incidence and risk factors. Phys Ther Sport. 2012 Nov;13(4):243-9. doi: 10.1016/j.ptsp.2012.01.001. Epub 2012 Feb 29. PMID 23068900